CLINICAL TRIAL: NCT07032220
Title: Application of Targeted Axillary Lymph Node Resection in Axillary Surgery After Neoadjuvant Chemotherapy for Breast Cancer: an Open-label, Multicenter Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chuan Wang, archiater, Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FujianUnions
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Surgery; Neoadjuvant Therapy; Sentinel Lymph Node Biopsy (SLNB)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and Accuracy of Targeted Axillary Dissection of Carbon Tattooing (Experimental)
  Interventions: Drug: carbon suspension

INTERVENTIONS:
Drug: carbon suspension — Before primary systemic therapy, a core needle biopsy or fine-needle aspiration of the most suspicious axillary lymph node was performed.22 Sterile black carbon suspension (0.5 mL: 25 mg, Chongqing LUMMY Pharmaceutical Co) was injected in the cortex of the metastatic node under ultrasound guidance using a 25G needle by a trained ultrasonographer at the time of biopsy or during a separate session. The injection volume was recorded and varied depending on node size and operator. The trained ultrasonographer had more than 5 years of puncture experience. Of note, for the patients with multiple abnormal nodes or N3 disease under ultrasound at diagnosis, only the pathologically-proven lymph node is marked with carbon suspension.

SUMMARY:
In this study, following the full informed consent of patients regarding the safety and potential benefits of the new intervention regimen, pathologically confirmed lymph nodes were pre-labeled with carbon nanoparticles prior to neoadjuvant chemotherapy. This was done to investigate the detection rate of carbon nanoparticle-labeled lymph nodes and to assess the stability and safety of carbon nanoparticles. Additionally, the dye single tracer method was employed for sentinel lymph node biopsy to evaluate the false-negative rate of TAD. This is an open-label, single-arm, multi-center prospective clinical trial. The primary objectives of this study are to evaluate the accuracy, feasibility, and safety of this method, thereby improving the quality of life and reducing postoperative complications for breast cancer patients while ensuring treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-70 years
2. The primary breast lesion was confirmed as invasive breast cancer by core needle biopsy
3. Axillary lymph node metastasis confirmed by fine needle aspiration or core needle biopsy
4. plan to undergo neoadjuvant chemotherapy
5. operable breast cancer
6. Patients with good heart, lung, liver, and kidney function are suitable for surgery
7. Informed consent

Exclusion Criteria:

1. Surgery is not planned or impossible
2. Metastasis of supraclavicular lymph nodes
3. distant metastasis, excluding bone metastasis
4. previous ipsilateral axillary surgery or radiotherapy
5. Due to personal or family factors, the patient is unable to cooperate with the surgical treatment recommended by the doctor according to the condition (breast conserving surgery or radical surgery).
6. Patients with severe heart and lung diseases, uncontrolled infectious diseases and other non-tumor related diseases could not tolerate comprehensive treatment such as surgery and chemotherapy
7. Unable to sign the informed consent form due to mental illness or other reasons
8. Poor medical compliance, and the study group believed that the patients could not complete the trial treatment process and follow-up according to the standard

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
By analyzing the detection rate of TAD, FNR and NPV, the feasibility and accuracy of this method in evaluating axillary lymph nodes of breast cancer patients after neoadjuvant therapy were evaluated. | 24 months

SECONDARY OUTCOMES:
The feasibility and accuracy of TLNB and SLNB in axillary lymph node evaluation were evaluated by analyzing the detection rate of TLNB and SLNB, FNR and NPV. | 24 months

OTHER OUTCOMES:
Evaluate the safety of carbon nanoparticles in breast cancer lymph node labeling | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Wang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Study Officials, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided